CLINICAL TRIAL: NCT01717040
Title: Double-Blind, Placebo-Controlled Trial of Pioglitazone for Bipolar Depression
Brief Title: Pioglitazone for the Treatment of Bipolar Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study ended early due to budgetary issues
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Joseph Calabrese, MD, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kemp DBDAT
Record Dates: First submitted 2012-04-17; First posted 2012-10-30 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: Bipolar Disorder; Insulin Resistance
Keywords: Bipolar Disorder; Insulin Resistance
MeSH Terms: conditions — Bipolar Disorder; Insulin Resistance | interventions — Pioglitazone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone will be initiated at a starting daily dose of 15 mg. After 7 days, the dose may be increased to 30 mg and after 35 days may be increased to a maximum of 45 mg per day.
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — Placebo will be initiated at a starting daily dose of 15 mg. After 7 days, the dose may be increased to 30 mg and after 35 days may be increased to a maximum of 45 mg per day.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The primary objective is to test the hypothesis that adjunctive pioglitazone is more effective than placebo for the relief of acute depressive symptoms resulting from bipolar disorder. The secondary objectives are to determine potential moderators and mediators of antidepressant efficacy.

DETAILED DESCRIPTION:
The study is a double-blind, placebo-controlled 8-week trial of pioglitazone, either as monotherapy or adjunctive to a mood stabilizer, for the acute relief of bipolar depression. The enrollment goal is 80 subjects (40 patients each in the pioglitazone treatment group and the placebo treatment group).

Screening Phase: Patients who have been prescribed a mood stabilizer for > 4 weeks and are on a therapeutic dose will proceed directly to the Screening Visit. For situations in which the patient prefers to be taking a mood stabilizer or where the treating psychiatrist feels it is clinically necessary, a mood stabilizer (lithium, divalproex, carbamazepine, lamotrigine, olanzapine, quetiapine, risperidone, aripiprazole, ziprasidone or lurasidone) will be initiated (see Mood Stabilizer Initiation section below). For this set of patients who do begin a mood stabilizer, the Screening Phase may last up to 8 weeks. Otherwise, subjects who do not come in on a mood stabilizer will proceed directly to screening.

Double-Blind, Placebo-Controlled Study Period (Week 1 to Week 8): Patients who meet inclusion/exclusion criteria will be randomized to study treatment at the baseline/randomization visit within 30 days of the screening visit. The efficacy and safety assessments will be carried out at baseline/randomization and then weekly or every two weeks for a total of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female >= 18 years of age
* Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis of bipolar disorder (type I, II, or NOS)
* Currently depressed as confirmed by the Mini-International Neuropsychiatric Interview (M.I.N.I.)-Plus at the screening visit
* Inventory of Depressive Symptoms total score > 25 or Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR16) > 11 at study baseline
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include barrier method with spermicide, abstinence, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.

Exclusion Criteria:

* Pregnant or breast feeding
* Unstable or inadequately treated medical illness as judged by the investigator
* Severe personality disorder
* Serious suicidal risk as judged by the investigator or having a score ≥ 4 on Montgomery Asberg Depression Rating Scale (MADRS) item number 10 (suicidal thoughts) at screening or baseline
* Known history of intolerance or hypersensitivity to pioglitazone
* Treatment with pioglitazone in the 3 months prior to randomization
* Dependence on alcohol or drugs (other than nicotine) in the 3 months prior to study entry
* Currently taking insulin or rosiglitazone.
* Diagnosed with dementia
* Acute Mania as defined by a Young Mania Rating Scale (YMRS) score > 15
* Diagnosed with heart failure
* Transaminase elevation >2.5 times the upper limit of normal
* Presence of renal impairment (eg. creatinine > 1.5)
* History of bladder carcinoma
* Fasting blood glucose >150 mg/dL and Hb A1c> 7%; participants meeting these criteria will be referred to an endocrinologist or their primary care physician for a diabetes evaluation and education.
* Receiving acute series of electroconvulsive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kemp, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center - Mood Disorders Program, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aftab A, Kemp DE, Ganocy SJ, Schinagle M, Conroy C, Brownrigg B, D'Arcangelo N, Goto T, Woods N, Serrano MB, Han H, Calabrese JR, Gao K. Double-blind, placebo-controlled trial of pioglitazone for bipolar depression. J Affect Disord. 2019 Feb 15;245:957-964. doi: 10.1016/j.jad.2018.11.090. Epub 2018 Nov 13. PMID 30699881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 17 | 20
Completed | 12 | 15
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Required Medication Change | 0 | 1
Not completed — New Substance Use Disorder | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.71 (12.071) | 43.65 (12.979) | 45.05 (12.492)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Bipolar Diagnosis [Count of Participants; unit: Participants]
  BP 1 | 11 | 13 | 24
  BP 2 | 5 | 7 | 12
  BP NOS | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) Total Score
Description: Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) is designed to assess the severity of depressive symptoms. Total scores can range from 0 to 84 with higher scores indicating a higher severity of depressive symptoms
Time Frame: Baseline and Week 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 17 | 20
units on a scale | 31.4 (3.0) | 24.3 (2.7)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 6/17 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=17) | Placebo (N=20)
Headache (General disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Confusion (General disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hot Flashes (General disorders) | 1 (1) | 0 (0)
Increased Urinary Frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shortness of Breath (Cardiac disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
Hair Loss (General disorders) | 0 (0) | 1 (1)
Increased Thirst (General disorders) | 0 (0) | 1 (1)
Stomach Upset (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tremor (General disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes